CLINICAL TRIAL: NCT01552070
Title: Impact of Alveolar Recruitment Maneuver on Extravascular Lung Water of Patients With Acute Lung Injury/Acute Respiratory Distress Syndrome.
Brief Title: Recruitment on Extravascular Lung Water in Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung Fu-Tsai, Chief of The Fifth Medical Intensive Care Unit , Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 99-0362A3
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With recruitment maneuver group (Experimental): Recruitment maneuver will be performed immediately (within 2 minutes) after intubation, consisting of a continuous positive airway pressure of 40 cmH2O over 30 seconds. Blood gases were sampled and blood samples taken for culture before, within 2 minutes, 5 minutes, and 30 minutes after intubation. Haemodynamic and respiratory parameters were continuously recorded throughout the study.
  Interventions: Behavioral: Recruitment maneuver
- Without recuritment maneuver (Active Comparator): After oral intubation, each patient will be mechanically ventilated, with a tidal volume of 6mL/kg, a respiratory rate of 20 to 25 breaths/minute, a positive end-expiratory pressure (PEEP) of 5 cmH2O, and an FiO2 of 100%. PEEP titration according to FiO2 and ARDSnet.
  Interventions: Other: without recruit maneuver

INTERVENTIONS:
Behavioral: Recruitment maneuver — Recruitment maneuver will be performed immediately (within 2 minutes) after intubation, consisting of a continuous positive airway pressure of 40 cmH2O over 30 seconds.
  Arms: With recruitment maneuver group
Other: without recruit maneuver — After oral intubation, each patient will be mechanically ventilated, with a tidal volume of 6mL/kg, a respiratory rate of 20 to 25 breaths/minute, a positive end-expiratory pressure (PEEP) of 5 cmH2O, and an FiO2 of 100%. PEEP titration according to FiO2 and ARDSnet.
  Arms: Without recuritment maneuver

SUMMARY:
The purpose of this study is to investigate the change of extravascular lung water (EVLW), cytokine and oxygenation parameters in patients with acute lung injury (ALI) or acute respiratory distress syndrome (ARDS) after alveolar recruitment maneuver.

DETAILED DESCRIPTION:
This investigation is a prospective randomized control study. Informed consents will be obtained from all patients or their surrogates prior to the procedure of alveolar recruitment maneuver and PiCCO monitoring system.

Patients and methods:

From September 2010 to September 2012, consecutive patients with ALI/ARDS undergo alveolar recruitment maneuver will be enrolled at Chang Gung Memorial Hospital, a university-affiliated hospital in Taiwan. EVLW will be measured by PiCCO monitoring system, alveolar recruitment maneuver will be setting by protocol under supervision of chest physicians and respiratory therapists. Serum cytokine such as endothelin-1, TNF-, IL-6, Tie-1, Tie-2, angiopoietin-1, angiopoietin-2,VEGF and thrombomodulin will be measured.

ELIGIBILITY:
Inclusion Criteria:

* acute hypoxemic respiratory failure requiring intubation; and hypoxemia, defined as a partial pressure of arterial oxygen (PaO2) less than 100 mmHg under a high fraction of inspired oxygen (FiO2)
* PaO2/FiO2 ratio < 200.

Exclusion Criteria:

* encephalopathy or coma,
* a need for cardiac resuscitation,
* hyperkalemia of more than 5.5 mEq/L (contraindication to the succinylcholine use),
* acute brain injury,
* pregnancy,
* age less 20 years old or recent thoracic surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Extravascular lung water change with/without recruitment maneuver. | 7 days
  The Extrvascular lung water (EVLW) measurement will be based on transpulmonary thermodilution method. This method was recently introduced as part of the PiCCO plus system (Pulsion Medical System, Munich, Germany). EVLW were recorded and compared between patients with and without recruitment manevuer.

SECONDARY OUTCOMES:
cytokines change with/without recruitment maneuver. | 28 days
  From September 2010 to September 2012, consecutive patients with ALI/ARDS undergo recruitment maneuver or not randomly will be enrolled. Serum cytokine such as endothelin-1, TNF-, IL-6, Tie-1, Tie-2, angiopoietin-1, angiopoietin-2,VEGF and thrombomodulin will be measured. Further ventilator use duration, weaning rate, ICU stay, safety and ICU survival were recorded and compared between patients with and without recruitment manevuer.
ventilator use duration | 28days
  From September 2010 to September 2012, consecutive patients with ALI/ARDS undergo recruitment maneuver or not randomly will be enrolled. Serum cytokine such as endothelin-1, TNF-, IL-6, Tie-1, Tie-2, angiopoietin-1, angiopoietin-2,VEGF and thrombomodulin will be measured. Further ventilator use duration, weaning rate, ICU stay, safety and ICU survival were recorded and compared between patients with and without recruitment manevuer.
weaning rate | 28days
  From September 2010 to September 2012, consecutive patients with ALI/ARDS undergo recruitment maneuver or not randomly will be enrolled. Serum cytokine such as endothelin-1, TNF-, IL-6, Tie-1, Tie-2, angiopoietin-1, angiopoietin-2,VEGF and thrombomodulin will be measured. Further ventilator use duration, weaning rate, ICU stay, safety and ICU survival were recorded and compared between patients with and without recruitment manevuer.
ICU stay | 28days
  From September 2010 to September 2012, consecutive patients with ALI/ARDS undergo recruitment maneuver or not randomly will be enrolled. Serum cytokine such as endothelin-1, TNF-, IL-6, Tie-1, Tie-2, angiopoietin-1, angiopoietin-2,VEGF and thrombomodulin will be measured. Further ventilator use duration, weaning rate, ICU stay, safety and ICU survival were recorded and compared between patients with and without recruitment manevuer.
ICU survival | 28days
  From September 2010 to September 2012, consecutive patients with ALI/ARDS undergo recruitment maneuver or not randomly will be enrolled. Serum cytokine such as endothelin-1, TNF-, IL-6, Tie-1, Tie-2, angiopoietin-1, angiopoietin-2,VEGF and thrombomodulin will be measured. Further ventilator use duration, weaning rate, ICU stay, safety and ICU survival were recorded and compared between patients with and without recruitment manevuer.

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Chyuan Lin, MD, Principal Investigator — Change Gung Memorial Hospital; Fu-Tsai Chung, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Department of Thoracic Medicine, Shuang Ho Hospital, Taipei Medical University, Taipei
  - Sant Paul Hospital, Taoyuan District